CLINICAL TRIAL: NCT07240896
Title: A Clinical Study on the Treatment of Wilson Disease With ATP7B mRNA/LNP (DSL101)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: DSciLab Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DSLIIT101
Record Dates: First submitted 2025-09-25; First posted 2025-11-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Wilsons Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: DSL101 (Experimental): Subjects will receive intravenous infusions of DSL101 once every four weeks.
  Interventions: Drug: Group 1: DSL101 Low dose
- Group 2: DSL101 (Experimental): Subjects will receive intravenous infusions of DSL101 once every four weeks.
  Interventions: Drug: Group 2: DSL101 Medium dose
- Group 3: DSL101 (Experimental): Subjects will receive intravenous infusions of DSL101 once every four weeks.
  Interventions: Drug: Group 3: DSL101 High dose

INTERVENTIONS:
Drug: Group 1: DSL101 Low dose — Subjects will receive intravenous infusions of DSL101 once every four weeks.
  Arms: Group 1: DSL101
Drug: Group 2: DSL101 Medium dose — Subjects will receive intravenous infusions of DSL101 once every four weeks.
  Arms: Group 2: DSL101
Drug: Group 3: DSL101 High dose — Subjects will receive intravenous infusions of DSL101 once every four weeks.
  Arms: Group 3: DSL101

SUMMARY:
This study adopted an open, single-arm, non-randomized, dose-escalation research design, aiming to evaluate the safety, tolerability, preliminary efficacy, pharmacokinetic and immunogenicity characteristics of single and multiple intravenous infusions of DSL101 in patients with Wilson's disease.

DETAILED DESCRIPTION:
In this study, low, medium and high dose groups were preset, the low dose group was accelerated titration group, and the medium and high dose groups used the traditional "3+3" method combined with Sentinel method for dose escalation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender not limited.
2. Meet the diagnostic criteria f Wilson's Disease in "Guidelines for Diagnosis and Treatment of Wilson's Disease (2022 Edition)", with a Leipzig score ≥4, at least one year between diagnosis and screening; ceruloplasmin level <0.1g/L.
3. Patinets with Wilson's disease confirmed by laboratory tests to have double-chromosome mutations in the ATP7B gene.
4. Low copper diet for at least six months befoer screening and willing to continue low copper diet during study.
5. Fertile subjects agreed to adopt reliable contrraceptive methods from the screening until 6 months after the last administration.
6. The subjects are atable patients with WD who have been trasted for at least six months without drug or dose changes for at least 6 momths at the time of screening , and have continuously used standard treatments [SOC, such as D-penicillamine, sodiu dihydroxypropane sulfonate, dimercaptosuccinic acid, trientine, and zinc preparations (zinc acetate, zinc gluconate, zinc sulfate)] for at least 6 months screening, and allowed subjects to continue with their prior SOC treatment.
7. The subject's condition was fully controlled after treatment, and its definition must meet all of the following conditions:

   1. Serum NCC level ≥ 25 μg/L and ≤ 150 μg/L;
   2. Urinary copper ≥100 μg/24 hours and ≤900 μg/24 hours;;
   3. ALT < 2 times of upper limit of normal value (ULN);
   4. The investigator believes that no other laboratory values or clinical symptoms would stop current standard therapy;
8. Subjects with good compliance, who can understand and cooperate to complete the requirements of protocol.
9. The subjects voluntarily participated in the trial and signed the informed consent form.

Exclusion Criteria:

1. Allergy or intolerance to the investigational drug.
2. Wilson's disease is accompanied by severe complications such as neurological and mental disorders.
3. History of liver transplantation.
4. Other liver-related diseases and clinical symptoms that can cause liver injury, such as acute and chronic hepatitis, alcoholic liver disease, autoimmune liver disease, drug-induced liver injury, liver cirrhosis, liver ascites, esophageal varices, hepatic encephalopathy, hepatorenal syndrome, liver failure, liver malignancy, etc.; Subjects with Model for end-stage liver disease score (MELD)>13.
5. Other diseases that can cause hemolysis or anemia, such as erythrocytosis, Mediterranean anemia, hemolytic anemia, various causes of infection, large area burns, etc.
6. Other diseases that can cause dysfunction of the nervous system, such as Parkinson's disease, Parkinson syndrome, various causes of dystonia, chorea, primary tremor, epilepsy, mental abnormalities (such as history of schizophrenia or suicide attempts), etc.
7. Screening period laboratory examination indicators:

   1. Hemoglobin < 90 g/L;
   2. Creatinine clearance ≤30 mL/min, or glomerular filtration rate <45 mL/min/1.73 m²;
   3. TBil≥2×ULN，ALP/TBil<4，AST/ALT>2.2;
   4. Platelets < 70 ×10^9/L;
   5. Neutrophils < 1.0 × 10^9 /L.
8. History of gastrointestinal bleeding within six months before screening.
9. Subjects with history of moderate to severe depression, suicidal thoughts or behaviors and serious psychiatric within 6 months prior to screening.
10. Subjects who have uncontrolled diseases of thr heart, liver, kidneys, endocrine system, digestive tract, metabolism, blood, or malignant tumors.
11. Active hepatitis B virus infection or active hepatitis C virus infection, or human immunodeficiency virus antibody positive.
12. Pregnant women or lactating women.
13. Subjects who have participated other clinical trial within 3 months prior to screening or plan to participate during the clinical trial.
14. Investigators evaluate other subjects who are not suitable to participate in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | up to 56 weeks

SECONDARY OUTCOMES:
Change in 24 hour urine copper | up to week 20
Change in sum total cpper [ serum copper bound by ceruloplasmin (NCC) ] | up to week 20
Change in serum free copper | up to week 20
Change from baseline in serum ceruloplasmin | up to week20
Change in serum iron concentration and serum ferritin concentration | up to week 20
Clinical laboratory test: Biochemistry - alanine aminotransferase (ALT) | up to week 20
  The physician will judge whether an abnormality is clinically significant
Change in the total score of the Unified Wilson Disease Rating Scale (UWDRS ) | up to week 20
  The UWDRS scale consists of three parts: neurological, liver function and mental symptom. The higher scores mean a worse outcome.
Number of subjects and percentage decrease in standard of care (SOC) medication euse within 20 weeks of administration | up to week 20
PK: Average steady-state concentration (Cav,ss) | up to week 6
Change from baseline in seurm ceruloplasmin activity | up to week20
Clinical laboratory test: Biochemistry - aspartate aminotransferase (AST) | up to week 20
Clinical laboratory test: Biochemistry - alkaline phosphatase (ALP) | up to week 20
Clinical laboratory test: Biochemistry - gamma-glutamyltransferase (γ-GGT) | up to week 20
Clinical laboratory test: Biochemistry - total bilirubin (TBIL) | up to week 20

OTHER OUTCOMES:
PK: Cmax | up to week 6
PK: Time to reach peak plasma concentration (Tmax) | up to week 6
PK: Area under the plasma concentration-time curve (AUC) | up to week 6
Immunogenicity: Positive rate of anti-drug antibody (ADA) | up to week 20

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
The study is in early stages and will consider releasing related information when sufficient data is available in subjects.